CLINICAL TRIAL: NCT01011426
Title: Bisacodyl Use in the Post-operative Care of Obstetrical/Gynecological (OB/GYN) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-148
Record Dates: First submitted 2009-11-07; First posted 2009-11-11 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Postoperative Nausea and Vomiting; Abdominal Pain
Keywords: laxative; postoperative care; ob-Gyn population; post-operative patients; obstetrical and gynecological surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Abdominal Pain | interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisacodyl (Active Comparator)
  Interventions: Drug: Bisacodyl
- empty opague capsule (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bisacodyl — 5mg po 6 hours postoperatively, repeat in 12 hours if no flatus
  Other Names: Dulcolax
  Arms: Bisacodyl
Drug: placebo — 1 capsule po 6 hours after surgery; repeat in 12 hours if no flatus
  Arms: empty opague capsule

SUMMARY:
The purpose of this study is to determine whether Bisacodyl, 5 mg usage decreases the incidence of nausea and abdominal pain after surgery, and also decreases the number of hospitalization days.

DETAILED DESCRIPTION:
Postoperative ileus is defined as a disturbance in bowel motility, clinically indistinguishable from bowel obstruction, and resulting from noxious or injurious bowel insult. During abdominal surgery, this could be due to bowel manipulation or its exposure to irritants like blood or pus. This contributes to post-operative morbidity resulting in significant patient discomfort and prolonged hospital stay. The clinical picture can be variable in presentation and severity. Patients can be asymptomatic or complain of anorexia, cramping, abdominal pain, nausea and vomiting, and bloating. Severe cases can have bilious vomiting. No diagnostic test can exclude the diagnosis with certainty and presence or absence of bowel sounds on exam is unreliable. Therefore, symptoms are primarily relied on for clinical management to promote patient comfort. Postoperative ileus can increase postoperative morbidity and lengthen hospital stay.

Traditionally, patients are given nothing-by-mouth (NPO) after major abdominal or pelvic surgery to allow rest for the dysfunctional bowel because of the concern of precipitating postoperative ileus. Patients are started on a clear liquid diet and advanced accordingly when there is documentation of bowel function such as passing flatus, presence of bowel sounds, or no obvious evidence of bowel obstruction such as nausea and vomiting. This was based on the fact that colonic motility is the last to recover after abdominal surgery (usually 3-5 days) and this is less precise in patients who develop constipation. However, the small bowel returns to normal peristaltic activity within 12-24 hours and the stomach within 24-48 hours. In addition, large body of evidence indicates that early feedings and early ambulation stimulates gastrointestinal motility, reduces overall complication rates as well as improves patient comfort and satisfaction. Laxatives also increase GI motility, will permit passage of flatus and/or stool, making the surgeon more comfortable in permitting early oral feeds. This will increase patient satisfaction, increase comfort by decreasing bloating and allow faster recovery. Bisacodyl is a mild laxative and so greatly suited for study in the post-operative period. However, laxative use can itself cause cramping, abdominal pain, and bloating.

There are several studies found in the literature about the effect of early bowel stimulation in postoperative care. However, there are only three studies related to the benefit of using laxatives during postoperative care to improve bowel function and decrease incidence of postoperative ileus. The Department of OB/GYN at Ohio showed earlier return to bowel function and a decrease in hospital stay while using Fleets Phosphorate Soda (66% sodium phosphate) in patients having a radical hysterectomy. Another study was done at Hvidovre University (Demark) to identify the benefit of using Magnesium Oxide and Disodium Phosphate immediately postoperatively in patients undergoing a hysterectomy. This study showed no difference on postoperative nausea, vomiting, or pain, but decreased the length of hospitalization by one day (N = 20). In July 2007, the Department of Surgery at Mahidol University (Thailand) used Bisacodyl suppositories on the third postoperative day in patients who underwent a colectomy for colon cancer. This study showed an increase incidence of postoperative ileus. All these studies are limited by their small number of patient enrollment, and none were blinded.

Bisacodyl (Dulcolax) is an over-the-counter laxative. It is coated with a protective coating so that it will not be digested in the stomach and small intestine. Therefore, Dulcolax only takes effect in the large intestine, where the coating is dissolved. Dulcolax is metabolized by the liver with CYP450 mechanism and excreted by stool and urine. Dulcolax works in the large intestine by stimulating the nerve endings, causing muscles to contract and the contents of the bowel to empty. Dulcolax is not used as the first treatment of bowel stimulation due to the concern about imbalance of electrolytes as well as dependency. There are few studies that document any adverse effect of Dulcolax. There are several studies showing Dulcolax as one the best choices of bowel prep agents without significant discomfort or imbalance of electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrical and gynecological patients undergoing abdominal surgery.

Exclusion Criteria:

* Subjects undergoing a bowel resection.
* Subjects who have a nasogastric tube for bowel decompression.
* Subjects allergic to Bisacodyl.
* Subjects with mechanical bowel obstruction undergoing bowel resection.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting in the 2 groups | 3-5 days

SECONDARY OUTCOMES:
Time to flatus | 2-5 days
Length of hospitalization | 2-5 days
Incidence of postoperative ileus | 2-5 days
Difference in pain scale in the 2 groups (Side-effects) | 2-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Meena Khandelwal, MD, Principal Investigator — Cooper University Hospital, NJ
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States